CLINICAL TRIAL: NCT01753362
Title: LIRAGLUTIDE IN OVERWEIGHT PATIENTS WITH TYPE 1 DIABETES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1965
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): subcutaneous daily injection
  Interventions: Drug: placebo
- liraglutide (Active Comparator): subcutaneous daily injection
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide
  Arms: liraglutide
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to examine the effects of liraglutide (a drug used to treat type 2 diabetes) on glucose (sugar) control over the 26 week study period when used in addition to insulin.

ELIGIBILITY:
Inclusion Criteria:

1) Type 1 Diabetes on continuous subcutaneous insulin infusion (CSII; also known as insulin pump) or multiple (four or more) injections of insulin per day. 2) Using a continuous glucose monitoring device (CGM) or regularly measuring their blood sugars four times daily. 3) HbA1c of less than 8.5%. 4) Well versed with carbohydrate counting. 5) Age 18-75 years 6) BMI≥ 25kg/m2 7) Age at diagnosis of type 1 diabetes should be <30 years. 8) evidence of auto-immunity to beta cells (GAD-65 and islet cell antibody screen)

Exclusion Criteria:

1)Type 1 diabetes for less than 6 months; 2)Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks; 3)Hepatic disease (transaminase > 3 times normal) or cirrhosis; 4)Renal impairment (serum eGFR <30ml/min/1.73m2); 5)HIV or Hepatitis B or C positive status; 6)Participation in any other concurrent clinical trial; 7)Any other life-threatening, non-cardiac disease; 8)Use of an investigational agent or therapeutic regimen within 30 days of study. 9) history of pancreatitis 10) pregnancy 11) inability to give informed consent 12) history of gastroparesis 13)history of medullary thyroid carcinoma or MEN 2 syndrome. 14) Smokers will be advised not to change their amount of smoking for the duration of the study; 15) Use of any agent other than insulin for treatment of diabetes (metformin, pramlintide or thiazolidinediones.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MBBS, Principal Investigator — SUNY UB
Locations (2):
- United States (2):
  - diabetes endocrinology center of WNY, Buffalo, New York
  - Diabetes Endocrinology Research Center of WNY, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: subcutaneous daily injection
  placebo
- Liraglutide: subcutaneous daily injection
  liraglutide
Period: Overall Study
Arm/Group | Placebo | Liraglutide
Started | 36 | 48
Completed | 26 | 40
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Liraglutide | Total
Number analyzed (Participants) | 26 | 40 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 36 | 58
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14.6) | 47 (13.0) | 47 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 42
  Male | 10 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 23 | 38 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 40 | 66

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: The primary endpoint of the study is to detect a difference in HbA1c percent at baseline and after 26 weeks of treatment with Liraglutide or placebo.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Placebo | Liraglutide
Number analyzed (Participants) | 26 | 40
percent
  baseline | 7.77 (0.83) | 7.94 (1.05)
  26 week | 7.64 (0.84) | 7.60 (0.98)

2. Secondary Outcome: Glucose Concentrations
Description: Mean daily glucose concentrations at baseline and 26 weeks
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Liraglutide
Number analyzed (Participants) | 26 | 40
mg/dL
  baseline | 183 (6) | 173 (8)
  26 week | 172 (5) | 171 (9)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Placebo | Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/40
Other Adverse Events (participants affected / at risk) | 0/26 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT01753362/Prot_SAP_000.pdf